CLINICAL TRIAL: NCT03283657
Title: Diabetes Risk Education and Communication Trial (DiRECT)
Brief Title: Diabetes Risk Education and Communication Trial
Acronym: DiRECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Matthew J O'Brien, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00204220; R34DK113541 (NIH)
Record Dates: First submitted 2017-08-22; First posted 2017-09-14 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: PreDiabetes; Diabetes Mellitus; Diabetes Mellitus, Type 2; Body Weight; Body Weight Changes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus; Diabetes Mellitus, Type 2; Body Weight; Body Weight Changes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DiRECT (Experimental): DiRECT consists of the following components that will be delivered by medical assistants before patients' routinely scheduled office visits: 1) a prediabetes decision aid focused on type 2 diabetes (T2D) risk and treatment options for preventing T2D; 2) a 'think aloud' exercise; and 3) formulating a preliminary treatment plan for T2D prevention.
  Interventions: Behavioral: DiRECT
- Usual Care (UC) (Active Comparator): Participants randomized to standard care will receive routine medical care without the medical assistant delivered DiRECT intervention.
  Interventions: Behavioral: Usual care (UC)

INTERVENTIONS:
Behavioral: DiRECT — DiRECT participants will meet with a medical assistant (MA) before a routinely scheduled office and formulate a preliminary treatment plan for T2D prevention. Participants will attend their scheduled physician visit, during which they may make a definitive treatment plan to initiate metformin and/or ILI.
  Arms: DiRECT
Behavioral: Usual care (UC) — Standard care with routine medical care.
  Arms: Usual Care (UC)

SUMMARY:
A large body of research has demonstrated that intensive lifestyle interventions and metformin are effective treatments to prevent or delay diabetes among high-risk adults, yet neither treatment is routinely used in practice. This pilot study will develop and evaluate the Diabetes Risk Education and Communication Trial (DiRECT) intervention, which communicates information about diabetes risk and treatment options for preventing diabetes among primary care patients with prediabetes. Given that 38% of U.S. adults have prediabetes, this project has large potential to impact public health by developing a scalable intervention to promote the use of evidence-based treatments that lower diabetes risk in this population.

DETAILED DESCRIPTION:
Landmark clinical trials have found that intensive lifestyle interventions (ILI) and metformin are safe and effective treatment options for preventing diabetes among adults with prediabetes and overweight/obesity. Despite being included in expert clinical guidelines, these treatments are rarely used in practice and little existing research has focused on approaches for promoting their use.

This novel intervention, delivered by medical assistants before patients' routinely scheduled office visits, consists of the following 3 components intended to promote initiation of ILI and metformin: 1) a prediabetes decision aid focused on diabetes risk and treatment options for preventing diabetes; 2) a "think aloud" exercise; and 3) formulating a preliminary treatment plan. Previous studies report that medical assistants can improve uptake of some preventive health services in primary care, which may also be true for ILI and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity
* documentation of prediabetes in medical chart or
* A1c 5.7-6.4

Exclusion Criteria:

* Age < 18; individuals who are not yet adults (infants, children, teenagers)
* Patient's primary care physician did not provide permission to participate in the study
* Pregnancy status: current or planned pregnancy during study period
* Serum creatinine >1.4mg/dL in women and >1.5mg/dL in men
* Patients that are blind, deaf, or otherwise unable to review study materials
* Prior diagnosis of diabetes mellitus type 1 or type 2 or on antidiabetic medication
* Diagnosis of post-surgical hypoinsulinemia
* Diagnosis of dementia
* Uncontrolled hypertension (≥160/100 mm Hg)
* No office visit in past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
Intent to treat questionnaire: Participant initiation of treatment to intensive lifestyle (ILI) or Metformin | 3 months
  The number of participants that initiate ILI, Metformin, or both treatments at follow-up is the primary outcome of the pilot trial, which will be assessed in the following ways. Because initiation of metformin requires a provider prescription, this will be assessed pragmatically using the electronic health record (EHR) and confirmed by participant self-report of taking at least 1 dose. Attendance logs will be used to confirm whether participants attended at least 1 ILI session. Those who received a prescription for metformin but do not take any doses will not be considered to have initiated treatment. Similarly, those who are referred to ILI but do not attend any sessions will not be classified as initiating treatment. Receiving a provider's prescription for metformin or referral for ILI without initiating treatment will be an exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J O'Brien, Principal Investigator — Assistant Professor
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Brien MJ, Cameron KA, Vargas MC, Mohr L, Williams GC, Fagerlin A, Kandula NR. Evaluation of a Prediabetes Decision Aid on Patient-Reported Outcomes in Primary Care: a Pilot Study. J Gen Intern Med. 2021 Mar;36(3):824-826. doi: 10.1007/s11606-020-05936-6. Epub 2020 Jun 15. No abstract available. PMID 32542497